CLINICAL TRIAL: NCT06823388
Title: Assessment of Acupuncture on Eye Fatigue : a Randomized Controlled Trial
Brief Title: Assessment of Acupuncture on Eye Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS1-24044
Record Dates: First submitted 2024-06-27; First posted 2025-02-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Acupuncture; Eye Fatigue; Accomodation
Keywords: eye fatigue; acupuncture
MeSH Terms: conditions — Asthenopia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Active Comparator)
  Interventions: Device: acupuncture
- pseudo-acupuncture group (Placebo Comparator)
  Interventions: Device: pseudo-acupuncture

INTERVENTIONS:
Device: acupuncture — acupuncture
  Arms: acupuncture group
Device: pseudo-acupuncture — The pseudo-acupuncture device can simulate the sensation of acupuncture stimulation.
  Arms: pseudo-acupuncture group

SUMMARY:
The study is designed to assess the effiacy of acupuncutre on eye fatigue. The indicator of eye fatigue is eye accommodation ability. Patients will be randomly assigned to the experimental group and the control group. The experimental group will receive acupuncture treatment, while the control group will receive sham acupuncture stimulation. The eye accommodation ability of both groups will be easured before and after the intervention, and the differences in eye accommodation ability before and after treatment will be analyzed.

DETAILED DESCRIPTION:
A dual-arm, parallel, randomized single-blind, sham-controlled trial will be conducted. The aim of the study is to assess the effiacy of acupuncutre on eye fatigue. Patients will be recruited from outpatient clinics. Subjects will be assessed at a Traditional Chinese Medicine (TCM) outpatient clinic and then have their accommodation function tested in an optometry room . This will determine if they meet the inclusion criteria.

Those who meet the inclusion criteria will be randomly assigned to the experimental group or the control group. The experimental group will receive treatment at seven acupuncture points: Fengfu (GV16), bilateral Fengchi (GB20), Yumen (TH2), and Hegu (LI4), using Jiasun 42G 1-inch acupuncture needles. The needles will be inserted perpendicularly to achieve the "De Qi" sensation, with a depth of 0.5 inches, and retained for 25 minutes before removal. The control group will undergo sham acupuncture at the same points using specially designed acupuncture needles from the manufacturer, which give the sensation of needling but retract into the handle without penetrating the skin, thus providing no real stimulation. Both groups will be treated by TCM physician .

After needle removal, visual acuity will be tested again to compare the differences in values between the pre- and post-test measurements of both groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjective experience of eye fatigue after using electronic devices at least twice a week.
* Age ≥ 18 years.
* Agreement to sign the informed consent form for this study.

Exclusion Criteria:

* Accommodation assessment: Interocular accommodation difference greater than 3 diopters (D).
* History of metabolic diseases with accompanying retinal conditions (e.g., diabetic retinopathy, hypertensive/hyperlipidemic patients with macular edema, retinal hemorrhage, glaucoma, etc.).
* Current treatment for ocular inflammation or infection (e.g., conjunctivitis, orbital cellulitis).
* Underwent eye surgery within the last 3 months (including LASIK surgery).
* Received acupuncture treatment for eye-related symptoms in the past month.
* Diagnosed with severe ophthalmic conditions (e.g., optic atrophy) and deemed unsuitable for the trial by an ophthalmologist.
* Diagnosed with anemia, hypotension, or chronic fatigue in the past three months, making them unsuitable for acupuncture due to a tendency to faint.
* Pregnant women.
* Major diseases such as renal insufficiency, cerebrovascular disease, or cancer, deemed unsuitable for clinical research participation by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
eye accommodation ability | From enrollment to the end of treatment in 30 minutes
  Value of eye accommodation ability difference before and after the intervention, measured by an autorefractor

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
eye accomodation ability